CLINICAL TRIAL: NCT04840524
Title: Effect of Preparation Design on the Functional and Esthetic Outcome of CAD/CAM Lithium Disilicate Laminate Veneers (Split Mouth Randomized Clinical Trial)
Brief Title: Effect of Preparation Design on the Functional and Esthetic Outcome of CAD/CAM Lithium Disilicate Laminate Veneers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Baher Ahmed Moustafa Ali, Assosiate lecturer of Fixed Prosthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-1-21; 20-1-21 (Registry Identifier: Research Ethics Committee)
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Dental Disorders Hard Tissues of Teeth; Tooth Discoloration
Keywords: Laminates; Vertical preparation; veneers
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional preparation design (Chamfer finish line with Butt joint incisal preparation design) (Other): conventional treatment
  Interventions: Procedure: Laminate veneers preparation
- New preparation design (Feather edge finish line with feather edge incisal preparation design) (Experimental): New preparation design
  Interventions: Procedure: Laminate veneers preparation

INTERVENTIONS:
Procedure: Laminate veneers preparation — facial laminate veneers teeth preparation

SUMMARY:
Conservatism is considered the main concern in any treatment plan, the feather edge preparation design of laminate veneers have been introduced yet clinical studies are lacking to evaluate their clinical performance.The aim of this study is to evaluate the effect of the two different preparation designs on the functional and esthetic outcome of laminate veneers in terms of marginal adaptation, retention, fracture, marginal discoloration and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* From 18-60 years old, and able to read and sign the informed consent document.
* Patients with teeth problems indicated for laminate veneers.
* Physically and psychologically able to tolerate conventional restorative procedures.
* Have no active periodontal or pulpal diseases.
* Maintenance of good oral hygiene .
* Willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth.
* Patients with para-functional habits.
* Cases that need modification in the incisal edge.
* Patients with poor oral hygiene and motivation .
* Psychiatric problems or unrealistic expectations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
marginal gap distance | at time of laminate cementation
  the gap between the laminate and the prepared tooth is measured before cementation using silicon replica and digital microscope

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No